CLINICAL TRIAL: NCT03913273
Title: Agonist-Antagonist Myoneural Interface for Functional Limb Restoration After Transtibial Amputation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts Institute of Technology (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1812634918; R01HD097135 (NIH)
Record Dates: First submitted 2019-04-11; First posted 2019-04-12 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Amputation
Keywords: Proprioception; Movement; Joint Prosthesis; Feedback; Rehabilitation

STUDY DESIGN:
Intervention Model Description: The study calls for an experimental group of eleven participants who underwent AMI transtibial amputations incorporating surgically constructed Agonist-antagonist Myoneural Interfaces (AMIs), and a control group of eleven participants who underwent standard transtibial amputations. Each participant in the control group is prospectively matched to a participant in the experimental group to the degree possible based on time since amputation, body habitus, age, and biological sex. Matching is conducted by methods that estimate causal effects by reducing imbalance in the matching variables; any differences in outcomes in the two groups should therefore be attributable to the AMIs. We anticipate that a planned number of thirty two enrolled, consented participants will allow us to account for participant attrition over time. The study protocol focuses on functional performance testing of a multi-degree of freedom prosthesis in fully healed participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention: AMI transtibial amputation
  Interventions: Procedure: AMI transtibial amputation
- Control group (Active Comparator): Intervention: Standard transtibial amputation
  Interventions: Procedure: Standard transtibial amputation

INTERVENTIONS:
Procedure: AMI transtibial amputation — Two Agonist-antagonist myoneural interfaces (AMIs) were surgically constructed during a modified transtibial amputation procedure. Each AMI was made of natively innervated and vascularized muscle segments - an agonist and antagonist - that were surgically connected in series within the amputated residuum. Tarsal tunnels, including segments of each tunnel's native tendon component, were procured from the amputated joint. The tunnels were affixed to the residual limb tibia and the AMIs were constructed by coaptation of an agonist and an antagonist muscle to either end of the tendon passing through the tunnel. Consequently, the force produced by one muscle stretches its partner such that the AMI can communicate signals from the mechanoreceptors in both muscles to the central nervous system.
  Arms: Intervention group
Procedure: Standard transtibial amputation — A standard transtibial amputation was performed according to traditional techniques. No surgical construction of agonist-antagonist myoneural interfaces (AMIs) was performed.
  Arms: Control group

SUMMARY:
This study involves the functional testing of a new lower extremity prosthesis by healthy, active participants with fully healed transtibial (below knee) amputations. The study design calls for an experimental group of eleven participants who received two agonist-antagonist myoneural interfaces (AMIs) that were surgically constructed during a modified transtibial amputation procedure, and a control group of eleven matched participants who received standard transtibial amputations. The study protocol involves one or more of the following activities:

1. Collection of electromyography (EMG) data from participants' lower limbs to characterize muscle activation and create maps specific to individual participants,
2. Investigation of participants' capabilities to use a new lower extremity prosthesis that is designed to allow independent actuation of the ankle and subtalar joints, and offers EMG-modulated control over prosthetic joint position and stiffness, and
3. Exploration of AMIs as a means of communicating information between the participant and the new prosthesis using an experimental system involving EMG, functional electrical stimulation, and ultrasound.

The hypothesis is that transtibial amputations involving AMIs can offer improved motor control of the new prosthesis while also enabling proprioceptive sensation (perception of the position, movement, and torque of the affected limb and prosthetic joint). The AMIs are expected to improve voluntary prosthetic control, improve prosthetic terrain adaptations, and offer new possibilities for bi-directional communication across the human-device interface.

DETAILED DESCRIPTION:
BACKGROUND:

Loss of limb profoundly impacts a person's health, productivity, independence, and quality of life. However, state-of-the-art medical and prosthesis technologies fall short of offering seamless human-device communication to those who require limb amputation. Ongoing, interactive efforts to advance amputation surgery techniques and develop novel "bionic" prostheses and prosthetic control systems are underway in an effort to address this interfacing challenge and thereby improve clinical outcomes within the population of amputees. We recently reported on the results of a first-in-human trial in which a prototype bionic prosthesis was tested in a recipient of a modified transtibial amputation. The modified amputation procedure involved the surgical construction of agonist-antagonist myoneural interfaces (AMIs) within the residual limb, where each AMI comprised two muscles - an agonist and an antagonist - connected in series. To enable the force produced by one muscle to cause stretch of its partner, "pulleys" were also constructed from the medial and lateral tarsal tunnels, including segments of each tunnel's native tendons, that were procured from the distal amputated limb and affixed to the residual limb tibia. The two AMIs were constructed via coaptation of the tibialis anterior and lateral gastrocnemius muscles to either end of the tendon portion passing through the proximally positioned tarsal tunnel, and coaptation of the tibialis posterior and peroneus longus muscles to either end of the tendon passing through the distally positioned tunnel. Following rehabilitation, this first recipient of the "AMI transtibial amputation" tested the feasibility of using his surgically constructed AMIs to control a prototype bionic prosthesis. The bionic prosthesis allowed motion in two degrees of freedom through independent actuation of powered ankle and subtalar joints, and the control algorithm allowed electromyography (EMG)-modulated control over prosthetic joint position and joint impedance.

Functional testing involved linking the proximal and distal AMIs within the participant's residual limb to the prosthetic ankle and subtalar joints through the use of surface EMG electrodes, intramuscular fine-wire electrodes, and functional electrical stimulation. The results of performance testing in this first AMI recipient suggested that AMIs can provide a biological tissue interface that can potentially offer a person with an amputation intuitive motor control of the affected limb and a bionic prosthesis while also enabling proprioception. The unique biomimetic tissue architecture of the AMI recapitulates a dynamic, mechanically functional muscle-tendon-muscle linkage that inherently provides mechanoreceptive biological sensors. Consequently, the AMI tissue architecture inherently preserves natural, bi-directional communication between surgically reconstructed limb musculature and the central nervous system, thereby building on and offering advantages over previously described neural interfacing approaches such as targeted muscle reinnervation (TMR), regenerative peripheral nerve interfaces (RPNIs), and peripheral nerve interfaces. Additionally, the surgical design implemented in the AMI transtibial amputation preserves the native innervation and vascularization for each nerve and muscle component, thereby offering a more robust, viable surgical construction than either TMR or RPNI, which instead rely upon the less robust regenerative processes of reinnervation and revascularization for long term viability. Long term functionality of the AMI is facilitated by the incorporation of autologous tarsal tendon and tunnel components, eliminating the need for either allogeneic grafts or synthetic implant materials. By providing a platform for robust efferent decoding of movement intent, as well as usable afferent feedback from a prosthetic joint, the AMI transtibial amputation paradigm has the potential to reinstate the human central nervous system as the primary mediator of prosthetic joint control.

STUDY OVERVIEW:

The goal of this clinical trial is to evaluate the efficacy of the AMI transtibial amputation.

STUDY POPULATION:

This study calls for healthy, active participants with transtibial amputations: an experimental group of participants who received AMI transtibial amputations, and a control group of participants who received standard transtibial amputations. Each participant in the control group is prospectively matched to a participant in the experimental group to the degree possible based on time since amputation, body habitus, age, and biological sex. We anticipate that a planned number of thirty-two enrolled, consented participants will allow us to account for participant attrition over time. As the population of lower limb amputees consists of participants of all genders and ethnicities, and since it is not practical to attempt to match all aspects of this variation in the context of a small study, this study aims to reflect the variation in the population of amputees to the degree possible.

EXPERIMENTAL SESSIONS:

Biomedical data are collected from study participants in the Biomechatronics space within the MIT Media Lab in Cambridge, MA. Experimental group participants attend five or six sessions, with four sessions lasting approximately 4 hours each and the other one or two session(s) lasting up to 8 hours. Control group participants attend four sessions lasting approximately 4 hours each.

HYPOTHESIS:

Surgically constructed AMIs within the amputated residuum can afford an improved independent control of joint position and impedance in a multi-degree-of-freedom prosthesis while also reflecting proprioceptive sensation from each prosthetic joint onto the central nervous system.

SPECIFIC AIM 1: Motion Control in Free Space

Aim 1 investigates if AMIs can improve voluntary free-space prosthetic control. Experimental and control group participants' capabilities for prosthetic control are evaluated and compared based on EMG and biomechanical measurements obtained during free-space voluntary movement tasks. In Aim 1A, data are collected using surface EMG sensors to characterize muscle activation, create maps specific to individual participants, and inform sensor requirements for subsequent aims. The data are obtained from a large number of EMG sensors that are distributed over participants' lower limbs. The participant is asked to move the phantom and/or biological foot through the ankle and subtalar joint spaces during data collection. Aim 1B explores if AMIs can improve motion control of a prosthesis that allows independent actuation of powered ankle and subtalar joint motions and EMG-modulated control over prosthetic joint positions and stiffnesses. Surface EMG data are obtained using a small number of sensors that are placed on participants' lower limbs at locations informed by the results of Aim 1A. Joint state data are collected from sensors on the prosthesis and other noninvasive sensors. Participants are asked to move their phantom ankle joints, in some cases mirroring specified motions of their unaffected limbs, in order to control the prosthesis. Performance tasks include pointing the prosthetic foot toward a specified position and stiffening the prosthetic joint to hold that position for a specified time interval.

SPECIFIC AIM 2: Terrain Adaptation

Aim 2 determines if AMIs can improve voluntary and involuntary (reflexive) prosthetic terrain adaptations. Experimental and control group participants' capabilities for prosthetic control are evaluated and compared based on EMG, biomechanical, and kinematic measurements that are obtained as they walk and traverse various terrains in a motion capture space. Surface EMG data are obtained using a small number of sensors that are placed on participants' lower limbs at locations informed by the results of Aim 1. Biomechanical data are collected from sensors on the prosthesis and sensors embedded in the terrain equipment. Kinematic data are collected wirelessly using a twelve-camera motion capture system. To facilitate kinematic data collection, reflective markers are affixed to the participant's clothes or skin to enable visualization and tracking of anatomical landmarks. Participants perform level ground walking and terrain adaptation tasks. One task involves navigating an obstacle presented in the participant's path during level ground walking. The task involves eversion of the prosthetic subtalar joint such that the lateral edge of the prosthetic foot contacts a vertically offset block while the medial edge of the prosthetic foot remains at the base height. Other tasks involve either descending or ascending stairs in sequential steps.

SPECIFIC AIM 3: Human-Device Communication

Aim 3 explores if AMIs can enable new possibilities for bi-directional human-device communication and provides data toward developing closed-loop prosthetic control strategies. Experimental group participants' capabilities to control prosthetic motion and their associated proprioceptive perceptions are investigated. EMG, ultrasound, biomechanical, and psychometric data are collected in the presence of varying levels of functional electrical stimulation (FES). The FES delivers a periodic stream of electrical pulses to target muscles in the participant's affected and unaffected limbs, causing contraction. One performance task involves an experimental pedal-pushing set-up. The participant is blindfolded and asked to plantar flex the phantom ankle joint, which causes the prosthetic ankle joint to press down on a foot pedal against mechanical resistance. Participants are also asked to plantar flex at varying effort levels and, in accordance with prosthetic sensor data resulting from each effort level, FES is applied to specific target muscles. Another task involves applying FES to specific target muscles in the affected limb and asking the participant to describe the perceived motions and forces and mirror these in the unaffected limb. In addition to participant responses, data are collected from fine-wire electrodes, surface EMG and other noninvasive sensors including an ultrasound imaging probe, and sensors on-board the prosthesis. Fine-wire FES and EMG electrodes are included in this study to reduce crosstalk that would interfere with the implementation of the prosthetic control strategy. The fine wire electrodes are placed by an experienced clinician in an acute setting; they do not remain in the limb. FES settings are kept within historically safe limits at all times. The FES begins at low intensity and is slowly increased until either the participant reports that a limit of comfortable stimulation has been reached or the historically safe limit is reached. The lower of these two values is established as a hard-stop reference for the FES setting.

ELIGIBILITY:
Inclusion Criteria:

Experimental group participants:

* Modified transtibial (below knee) amputation incorporating agonist-antagonist myoneural interfaces (AMIs) and performed at the Brigham and Women's Hospital, Boston, MA.
* Fully healed amputation site
* Proficiency in using a standard lower extremity prosthesis
* Activity or K-Level of at least K3 to K4 (capability to ambulate with variable cadence)

Control group participants:

* Standard transtibial (below knee) amputation
* Fully healed amputation site
* Proficiency in using a standard lower extremity prosthesis
* Activity or K-Level of at least K3 to K4 (capability to ambulate with variable cadence)

Exclusion Criteria

Experimental and Control group participants:

* Persons beyond the stated age restrictions
* Persons with one or more of the following underlying health conditions: cardiopulmonary instability manifest as coronary artery disease, chronic obstructive pulmonary disease, and extensive microvascular compromise
* Persons who are active smokers
* Persons who are pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-06-12 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Stability of Joint Position Control in Free Space | 0 - 5 years
  A measure of the capability to maintain prosthetic joint position in free space. Determined as the amount of time the prosthesis can be maintained in a given position relative to the requested hold time.
Economy of Motion during Joint Position and Impedance Control in Free Space | 0 - 5 years
  A measure of the distance traversed by the prosthetic joint during a target tracking task involving position and impedance control in free space. Determined as the total travel distance, in angle space, normalized by the minimum travel distance from start to finish.
Subtalar Eversion for an Obstacle | 0 - 5 years
  A measure of the capability to navigate an obstacle presented in the participant's path. The task involves eversion of the prosthetic subtalar joint such that the lateral edge of the prosthetic foot contacts a vertically offset block while the medial edge of the prosthetic foot remains at the base height. Determined as the maximum late-swing subtalar joint eversion angle measured between 80 and 100 percent of the participant's gait cycle during task performance.
Late Swing Ankle Plantar Flexion during Stair Descent | 0 - 5 years
  A measure of the capability to exhibit prosthetic ankle joint plantar flexion that is characteristic of stair descent. Determined as the maximum late-swing ankle joint plantar flexion angle measured between 80 and 100 percent of the participant's gait cycle during task performance.
Late Swing Ankle Dorsiflexion during Stair Ascent | 0 - 5 years
  A measure of the capability to exhibit prosthetic ankle joint dorsiflexion that is characteristic of stair ascent. Determined as the maximum late-swing ankle joint dorsiflexion angle measured between 80 and 100 percent of the participant's gait cycle during task performance.

SECONDARY OUTCOMES:
Correlation and Repeatability of Ankle Joint Proprioception | 0 - 5 years
  A measure of the correlation of force estimated within the agonist-antagonist muscle unit with the participant's reported perception of prosthetic joint torque.
Controllability over Prosthetic Joint Plantar Flexion Torque | 0 - 5 years
  A measure of the number of participant plantar flexion effort levels that resulted in torque production that differed significantly from the torques produced at all other effort levels.

CONTACTS AND LOCATIONS:
Overall Officials: Hugh M Herr, PhD, Principal Investigator — Massachusetts Institute of Technology
Locations (1):
- Massachusetts Institute of Technology, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Srinivasan SS, Carty MJ, Calvaresi PW, Clites TR, Maimon BE, Taylor CR, Zorzos AN, Herr H. On prosthetic control: A regenerative agonist-antagonist myoneural interface. Sci Robot. 2017 May 31;2(6):eaan2971. doi: 10.1126/scirobotics.aan2971. PMID 33157872
- [Background] Clites TR, Carty MJ, Ullauri JB, Carney ME, Mooney LM, Duval JF, Srinivasan SS, Herr HM. Proprioception from a neurally controlled lower-extremity prosthesis. Sci Transl Med. 2018 May 30;10(443):eaap8373. doi: 10.1126/scitranslmed.aap8373. PMID 29848665
- [Background] Clites TR, Herr HM, Srinivasan SS, Zorzos AN, Carty MJ. The Ewing Amputation: The First Human Implementation of the Agonist-Antagonist Myoneural Interface. Plast Reconstr Surg Glob Open. 2018 Nov 16;6(11):e1997. doi: 10.1097/GOX.0000000000001997. eCollection 2018 Nov. PMID 30881798
- [Background] Amtmann D, Morgan SJ, Kim J, Hafner BJ. Health-related profiles of people with lower limb loss. Arch Phys Med Rehabil. 2015 Aug;96(8):1474-83. doi: 10.1016/j.apmr.2015.03.024. Epub 2015 Apr 25. PMID 25917819
- [Background] Kurichi JE, Vogel WB, Kwong PL, Xie D, Bates BE, Stineman MG. Factors associated with total inpatient costs and length of stay during surgical hospitalization among veterans who underwent lower extremity amputation. Am J Phys Med Rehabil. 2013 Mar;92(3):203-14. doi: 10.1097/PHM.0b013e31827446eb. PMID 23117271
- [Background] Ziegler-Graham K, MacKenzie EJ, Ephraim PL, Travison TG, Brookmeyer R. Estimating the prevalence of limb loss in the United States: 2005 to 2050. Arch Phys Med Rehabil. 2008 Mar;89(3):422-9. doi: 10.1016/j.apmr.2007.11.005. PMID 18295618
- [Background] Herr HM, Grabowski AM. Bionic ankle-foot prosthesis normalizes walking gait for persons with leg amputation. Proc Biol Sci. 2012 Feb 7;279(1728):457-64. doi: 10.1098/rspb.2011.1194. Epub 2011 Jul 13. PMID 21752817
- [Background] Stolyarov R, Burnett G, Herr H. Translational Motion Tracking of Leg Joints for Enhanced Prediction of Walking Tasks. IEEE Trans Biomed Eng. 2018 Apr;65(4):763-769. doi: 10.1109/TBME.2017.2718528. Epub 2017 Jun 22. PMID 28650802
- [Background] Huang S, Huang H. Voluntary Control of Residual Antagonistic Muscles in Transtibial Amputees: Reciprocal Activation, Coactivation, and Implications for Direct Neural Control of Powered Lower Limb Prostheses. IEEE Trans Neural Syst Rehabil Eng. 2019 Jan;27(1):85-95. doi: 10.1109/TNSRE.2018.2885641. Epub 2018 Dec 7. PMID 30530332
- [Background] Hargrove LJ, Simon AM, Young AJ, Lipschutz RD, Finucane SB, Smith DG, Kuiken TA. Robotic leg control with EMG decoding in an amputee with nerve transfers. N Engl J Med. 2013 Sep 26;369(13):1237-42. doi: 10.1056/NEJMoa1300126. PMID 24066744
- [Background] Irwin ZT, Schroeder KE, Vu PP, Tat DM, Bullard AJ, Woo SL, Sando IC, Urbanchek MG, Cederna PS, Chestek CA. Chronic recording of hand prosthesis control signals via a regenerative peripheral nerve interface in a rhesus macaque. J Neural Eng. 2016 Aug;13(4):046007. doi: 10.1088/1741-2560/13/4/046007. Epub 2016 Jun 1. PMID 27247270
- [Background] Ortiz-Catalan M, Hakansson B, Branemark R. An osseointegrated human-machine gateway for long-term sensory feedback and motor control of artificial limbs. Sci Transl Med. 2014 Oct 8;6(257):257re6. doi: 10.1126/scitranslmed.3008933. PMID 25298322
- [Background] Schiefer M, Tan D, Sidek SM, Tyler DJ. Sensory feedback by peripheral nerve stimulation improves task performance in individuals with upper limb loss using a myoelectric prosthesis. J Neural Eng. 2016 Feb;13(1):016001. doi: 10.1088/1741-2560/13/1/016001. Epub 2015 Dec 8. PMID 26643802
- [Derived] Srinivasan SS, Gutierrez-Arango S, Teng AC, Israel E, Song H, Bailey ZK, Carty MJ, Freed LE, Herr HM. Neural interfacing architecture enables enhanced motor control and residual limb functionality postamputation. Proc Natl Acad Sci U S A. 2021 Mar 2;118(9):e2019555118. doi: 10.1073/pnas.2019555118. PMID 33593940
- See also: STAT Documentary on the "Ewing" amputation surgery — https://www.statnews.com/2018/05/30/pioneering-amputation-surgery-prosthetic-foot/
- See also: Brigham and Women's hospital video on the "Ewing" amputation surgery — https://www.brighamandwomensfaulkner.org/about-bwfh/news/ewing